CLINICAL TRIAL: NCT05820841
Title: A Randomized, Open-label, Phase 3 Study of Acalabrutinib in Combination With Rituximab and Reduced Dose CHOP (R-miniCHOP) in OldEr Adults With Untreated Diffuse Large B-Cell Lymphoma
Brief Title: Acalabrutinib in Combination With R-miniCHOP in Older Adults With Untreated Diffuse Large B-Cell Lymphoma
Acronym: ARCHED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Collaborators: University of Leipzig (Other); University Hospital Regensburg (Other); Wuerzburg University Hospital (Other); University Hospital of Gießen and Marburg (Unknown); Saarland University Medical Center (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARCHED / GLA 2022-1; U1111-1284-7084 (Other: WHO - Universal Trial Number); 2022-501187-18-00 (Other: EU Clinical Trial Number:)
Record Dates: First submitted 2023-03-08; First posted 2023-04-20 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Large B-cell Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: Diffuse large B cell lymphoma; Older adults; Geriatric; Large B cell lymphoma; Aggressive B cell lymphoma; Acalabrutinib; R-miniCHOP; R-mini-CHOP; BTK inhibitor
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard arm (Active Comparator): 6x R-miniCHOP + 2x Rituximab.
  Interventions: Drug: R-miniCHOP
- Experimental arm (Experimental): 6x R-miniCHOP + 2x Rituximab + Acalabrutinib.
  Interventions: Drug: R-miniCHOP + Acalabrutinib

INTERVENTIONS:
Drug: R-miniCHOP + Acalabrutinib — * Rituximab i.v.: 375 mg/m2 (D0)
  * Cyclophosphamide i.v.: 400 mg/m² (D1)
  * Doxorubicin i.v.: 25 mg/m² (D1)
  * Vincristine i.v.: 1 mg (D1)
  * Prednisolone p.o.: 40 mg/m² (D1 to D5)
  * Acalabrutinib 100 mg p.o. twice daily starting from D1 of first R-miniCHOP cycle continuously to D21 of cycle 8.
  Cycles repeated every 3 weeks
  Arms: Experimental arm
Drug: R-miniCHOP — * Rituximab i.v.: 375 mg/m2 (D0)
  * Cyclophosphamide i.v.: 400 mg/m² (D1)
  * Doxorubicin i.v.: 25 mg/m² (D1)
  * Vincristine i.v.: 1 mg (D1)
  * Prednisolone p.o.: 40 mg/m² (D1 to D5).
  Cycles repeated every 3 weeks
  Arms: Standard arm

SUMMARY:
The goal of this clinical trial is to study the addition of Acalabrutinib to standard R-miniCHOP in older adults with DLBCL. The main question it aims to answer is whether progression free survival kann be prolonged with the addition of Acalabrutinib.

Participants will be randomised to receive either R-miniCHOP alone or R-miniCHOP with Acalabrutinib.

ELIGIBILITY:
Inclusion Criteria:

Informed consent

1. Ability to understand the purpose and risks of the study and capable of giving signed informed consent which includes:

   1. Compliance with the requirements and restrictions listed in the informed consent form (ICF).
   2. Authorization to use protected health information/data [in accordance with the General Data Protection Regulation (GDPR)].
2. Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses
3. Willing and able to participate in all required evaluations and procedures in this study protocol, including swallowing capsules and tablets without difficulty.

   Age/Sex
4. Men and women >80 years of age or >60 up to 80 years of age and ineligible for full dose R-CHOP according to investigator assessment*.

   We recommend classifying patients aged 61-80 as full-dose R-CHOP ineligible if they fulfill one of the following criteria: ADL <5, IADL <6, CIRS-G ≥1 score = 3, or > 8 score = 2.
5. Male patients who are sexually active with women of childbearing potential (definitions see section 17.8) must agree to use highly effective forms of contraception with the addition of a barrier method (condom) during the study (see section 17.8.1) as well as to the restrictions mentioned in section 9.13.
6. Female patients of childbearing potential (definitions see 17.8) who are sexually active must agree to use highly effective forms of contraception while on the study as well as to the restrictions mentioned in section 9.13.

   Disease characteristics
7. Histologically proven, previously untreated CD20+ diffuse large B-cell lymphoma (DLBCL) according to the 2017 WHO classification including:

   1. diffuse large B-cell lymphoma (DLBCL), not otherwise specified (NOS)
   2. primary cutaneous DLBCL leg type
   3. intravascular large B-cell lymphoma
   4. EBV+ DLBCL, NOS
   5. HHV8+DLBCL, NOS
   6. primary mediastinal (thymic) large B-cell lymphoma
   7. B-cell lymphoma, with intermediate features between DLBCL and classical Hodgkin lymphoma
   8. follicular lymphoma grade 3B
   9. high-grade B-cell lymphoma, NOS
   10. high-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements
   11. T-cell/histiocyte-rich large B-cell lymphoma
   12. DLBCL associated with chronic inflammation
   13. ALK+ large B-cell lymphoma
   14. large B-cell lymphoma with IRF4 rearrangement Please note: patients in whom indolent lymphoma is diagnosed concurrently with the one of the above listed diagnoses can also be included.
8. Disease Stage I with bulk ≥7.5cm, II, III or IV according to Ann Arbor Classification Type of patient and clinical characteristics
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2. An ECOG Score of 3 is acceptable only if this is directly attributable to lymphoma.
10. Meet the following laboratory parameters:

    1. Absolute neutrophil count (ANC) ≥ 1500 cells/µl or platelet count ≥ 100.000/µl unless directly attributable to lymphoma.
    2. Serum AST and ALT ≤3 x upper limit of normal (ULN) unless directly attributable to lymphoma.
    3. Total bilirubin ≤1.5 x ULN, unless directly attributable to Gilbert's syndrome or lymphoma.
    4. Estimated creatinine clearance of ≥30 mL/min, calculated by Cockcroft-Gault (using actual body weight) (if male, [140-Age] x Mass [kg] / [72 x creatinine mg/dL]; multiply by 0.85 if female), or serum creatinine ≤2.5 x ULN.

Exclusion Criteria:

Medical conditions

1. Evidence of disease (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension and renal transplant) that, in the investigator's opinion, make it undesirable for the patient to participate in the study or that would jeopardize compliance with the protocol [e.g. a single score of 4 on one single category on the CIRS-G-Score (but not a cumulative score of 4)].
2. Significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of randomization or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or LVEF < 40%. Patients with controlled, asymptomatic atrial fibrillation are allowed to enroll on study.
3. Severe pulmonary dysfunction (CTCAE grade 3 or 4) unless associated with lymphoma.
4. Severe psychiatric or neurologic disease that, in the investigator's opinion, make it undesirable for the patient to participate in the study or that would jeopardize compliance with the protocol.
5. Persistent neuropathy CTCAE grade 3 or 4.
6. Refractory nausea and vomiting, inability to swallow acalabrutinib, or malabsorption syndrome; chronic severe gastrointestinal disease, gastric restrictions, or bariatric surgery such as gastric bypass; partial or complete bowel obstruction, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of study treatment.
7. History of prior malignancy that could affect compliance with the protocol or interpretation of results, except for the following:

   1. Curatively treated localised basal cell carcinoma or localised squamous cell carcinoma of the skin or carcinoma in situ of the cervix or carcinoma in situ / low risk carcinoma of the prostate requiring only observation, as well as untreated low grade lymphoma except chronic lymphocytic leukemia.
   2. Other cancers not specified above that have been curatively treated by surgery and/or radiation therapy from which patient is disease-free for ≥2 years (≥5 years for those treated with chemotherapy) without further treatment or which are not expected to limit survival to < 2 years.
8. Received a live virus vaccination within 28 days of randomization.
9. Known history of infection with HIV.
10. Any active significant infection (e.g., bacterial, viral or fungal) as assessed by the investigator.
11. History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML).
12. Serologic status reflecting active hepatitis B or C infection.

    1. Patients who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative PCR result before randomization and must be willing to undergo DNA PCR testing during the study. Those who are HBsAg-positive or hepatitis B PCR positive will be excluded.
    2. Patients who are hepatitis C antibody positive will need to have a negative PCR result before randomization. Those who are hepatitis C PCR positive will be excluded.
13. History of stroke or intracranial hemorrhage within 6 months before randomization.
14. History of clinically relevant bleeding diathesis (e.g., hemophilia, von Willebrand disease).
15. Major surgical procedure within 30 days before randomization. Note: If a patient had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
16. Breastfeeding or pregnant women.
17. Current life-threatening illness, medical condition, organ system dysfunction, social, geographical or economic condition which, in the Investigator's opinion, could compromise the patient's safety or put the study at risk.
18. Diagnosis of primary central nervous system lymphoma or secondary central nervous system or meningeal involvement by lymphoma
19. Diagnosis of Richter's Transformation/transformed CLL Prior/Concomitant therapy
20. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists. Patients using therapeutic low molecule weight heparin, direct oral anticoagulants or low dose aspirin will be eligible. Switching from vitamin K antagonists to one of the allowed anticoagulants above prior to trial entry is permitted.
21. Requires treatment with a strong cytochrome P450 3A (CYP3A) inhibitor or inducer. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study drug is prohibited. See details in section 9.12.1.
22. Prior exposure to a BTK inhibitor.
23. Prior anthracycline use ≥300 mg/m2.
24. Already initiated lymphoma therapy except for steroid (max. total dose of 1000mg), vincristine (max. 1 mg once) or rituximab (max. 375mg/m2) prephase.
25. Concurrent participation in another therapeutic clinical trial.
26. Requires treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Patients receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrolment into this study.
27. Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug.

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) investigator assessed | Up to 5 years
  PFS, defined by the time between the day of randomization until one of the following events occurs, whichever comes first: Disease progression (PD), relapse after complete remission (CR) or death due to any cause, as per Lugano Classification of 2014. Patients who have not experienced an event at the time of analysis will be censored at the most recent date of disease assessment.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  OS, defined by the time between the day of randomization until death due to any cause. Patients who have not experienced an event at the time of analysis will be censored at the date when the patient was last known to be alive.
PFS based on blinded independent central review (BICR) | Up to 5 years
Event-free survival (EFS) | Up to 5 years
  EFS, defined by the time between the day of randomization until one of the following events occurs, whichever comes first: Progressive disease (PD), relapse after complete remission (CR), initiation of subsequent systemic anti-lymphoma treatment and/or irradiation or death due to any cause, as per Lugano Classification of 2014.
PFS according to Cell of Origin as per immunohistochemistry | Up to 5 years
OS according to Cell of Origin as per immunohistochemistry | Up to 5 years
EFS according to Cell of Origin as per immunohistochemistry | Up to 5 years
PFS according to molecular genotype | Up to 5 years
OS according to molecular genotype | Up to 5 years
EFS according to molecular genotype | Up to 5 years
Complete (CR) partial (PR) and overall (ORR) remission rates | Up to 5 years
Duration of Response (DoR) | Up to 5 years
Progression rate, relapse rate and central nervous system (CNS) relapse rate | Up to 5 years
Adverse events (AEs), Serious AEs, AEs of special interest, events of clinical interest, AEs leading to study treatment discontinuation or dose modification. | Up to 5 years
Rate of secondary malignancies | Up to 5 years
Treatment-related death rate | Up to 5 years
Dose intensity of miniCHOP, rituximab and acalabrutinib. | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Christofyllakis, MD MSc, Principal Investigator — Saarland University Medical Center; Moritz Bewarder, MD, PD, Principal Investigator — Saarland University Medical Center
Locations (17):
- Germany (17):
  - Saarland University Medical Center, Homburg, Saarland
  - MVZ am Klinikum Aschaffenburg, Aschaffenburg
  - Helios Klinikum Emil von Behring, Berlin
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Gemeinschaftspraxis Mohm/Prange-Krex, Dresden
  - Universitätsklinikum Gießen und Marburg, Standort Gießen, Giessen
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsmedizin Halle (Saale), Halle
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Johannes Wesling Klinikum, Minden
  - Rheinland Klinikum-Lukaskrankenhaus Neuss, Neuss
  - Brüderkrankenhaus St. Josef, Paderborn
  - CaritasKlinikum Saarbrücken St. Theresia, Saarbrücken
  - Klinikum Mutterhaus der Borromäerinnen, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Bundeswehrkrankenhaus Ulm, Ulm
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided